CLINICAL TRIAL: NCT04970095
Title: Evaluation of Alt-RAMEC by EDO With Facemask in Patients With Cleft Lip and Palate (UCLP) Using Cone Beam Computed Tomography (CBCT)
Brief Title: Alt-RAMEC Expansion and Protraction by EDO in Cleft Lip and Palate Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, sarah salah khalil Abdelaal, Principal Investigator, Faculty of Dental Medicine for Girls
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORTHO-109-2-F
Record Dates: First submitted 2021-07-16; First posted 2021-07-21 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Cleft Lip and Palate
Keywords: Alt-RAMEC; expansion; cleft lip and palate patient; cone beam computed tomography (CBCT); protraction; facemask; MAXILLARY EXPANDER WITH DIFFERENTIAL OPENING (EDO)
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cleft lip and palate patient (Experimental): Clefts patient with transverse maxillary constriction and anteroposterior deficiency
  Interventions: Device: Maxillary Expander with Differential Opening (EDO); Device: Petit Face Mask

INTERVENTIONS:
Device: Maxillary Expander with Differential Opening (EDO) — The EDO is designed with two expansion screws positioned transversely. When more expansion is required between the canines, the anterior screw can be further activated. Both expansion screws can be activated to open in a parallel configuration. Pivoting corner screws allow for different amounts of expansion without significant risk of binding during activation.
Device: Petit Face Mask — The face mask is anatomical, multi-adjustable, lightweight and an ideal therapeutic alternative for the correction of Class III malocclusion.
  consist of forehead cap chin cap cross bar

SUMMARY:
Evaluate the treatment outcome of Alternate Rapid Maxillary Expansion and Constriction Alt-RAMEC protocol on patients with cleft lip and palate, using a differential opening expander and face mask which will be measured and recorded by cone beam computed tomography (CBCT).

DETAILED DESCRIPTION:
Cleft lip and palate are among the most common deformities in children.Clefts patient are usually having orofacial problems as missing or unerupted permanent teeth, alveolar bone defect, speech difficulty . Patients with cleft lip and palate (CLP) commonly have maxillary arch constriction (maxillary hypoplasia) and Class III malocclusions due to deficient of maxillary growth The upper jaw of patients with cleft palate will be expanded by Maxillary Expander with Differential Opening (EDO) with alternate rapid maxillary expansion and constriction (Alt-RAMEC) , which is opened by opening the expansion device by 1 mm per day for a week, then closing the device at a rate of 1 mm per day in the second week and so on alternately for 7 consecutive weeks after the completion of the expansion, the facemask device will be used to protraction of maxilla the measurement and difference before and after treatment will be assessment by cone beam computed tomography (CBCT). .

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Cleft lip and palate patients.
* All patient age ranges from 8 to 12 years.
* All the cases showed maxillary arch constriction and deficiently
* All patients had maxillary permanent first molars.
* Primary lip adhesion and palatal closure.

Exclusion Criteria:

* Patients had received any surgical assisted expansion or maxillary protraction or fixed orthodontics before.

  2. Maxillary dentition unsuitable to bond the expander (less than two dental unit bedside first permanent molar) .

  3. Absent maxillary permanent first molars. 4. Uncooperative patients/parents

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
change in 3D dimension of skull after and before expansion | six month
  Full skull Cone Beam Computerized Tomography

CONTACTS AND LOCATIONS:
Overall Officials: maha m. mohamed, phd, Study Director — Lecturer of Orthodontics Department Faculty of Dental Medicine for Girls Al-Azhar University
Locations (1):
- faculty of dental medicine for Girls, Al- Azhar University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No
Evaluation of EDO ,Alt-RAMEC With Facemask in Patients With Cleft lip and Palate (UCLP) Using Cone Beam Computed Tomography (CBCT)

REFERENCES:
- [Background] Garib D, Lauris RC, Calil LR, Alves AC, Janson G, De Almeida AM, Cevidanes LH, Lauris JR. Dentoskeletal outcomes of a rapid maxillary expander with differential opening in patients with bilateral cleft lip and palate: A prospective clinical trial. Am J Orthod Dentofacial Orthop. 2016 Oct;150(4):564-574. doi: 10.1016/j.ajodo.2016.05.006. PMID 27692413
- [Background] Singh S, Batra P, Raghavan S, Sharma K, Srivastava A. Evaluation of Alt-RAMEC With Facemask in Patients With Unilateral Cleft lip and Palate (UCLP) Using Cone Beam Computed Tomography (CBCT) and Finite Element Modeling-A Clinical Prospective Study. Cleft Palate Craniofac J. 2022 Feb;59(2):166-176. doi: 10.1177/10556656211000968. Epub 2021 Mar 23. PMID 33754882
- See also: Maxillary Expander with Differential Opening (EDO) — https://www.greatlakesdentaltech.com/maxillary-expander-with-differential-opening-edo.html